CLINICAL TRIAL: NCT07212517
Title: The Effect of Benson Relaxation Exercises on Sleep Quality in Patients With Lung Cancer
Brief Title: Benson Relaxation Exercises and Sleep Quality in Lung Cancer Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, elçin babaoğlu, Asst. Dr. (Psychiatric Nursing), Uskudar University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: UU-NURSE-RK-04
Record Dates: First submitted 2025-09-30; First posted 2025-10-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-09

CONDITIONS: Sleep Quality; Relaxation; Canser; Benson Exercise
Keywords: cancer patient; Benson relaxation; sleep Quality
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: randomized controlled trial single blinded
Who Masked: Participant
Masking Description: experimental and control groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): patients will be randomly assigned to groups using this program. Patients included in the study will be numbered according to their order of arrival and assigned to the intervention and control groups according to the order in the randomization listThis study is planned to be conducted on patients diagnosed with lung disease. Patients with additional mental illness, oxygen saturation values below 90, pain scores above 5, and bloody sputum will be excluded from the study.
  Interventions: Behavioral: benson relaxation exercise
- control (No Intervention): Patients will be randomly assigned to groups using this program. Patients included in the study will be numbered according to their order of arrival and assigned to the intervention and control groups according to the order in the randomization listThis study is planned to be conducted on patients diagnosed with lung disease. Patients with additional mental illness, oxygen saturation values below 90, pain scores above 5, and bloody sputum will be excluded from the study.

INTERVENTIONS:
Behavioral: benson relaxation exercise — BRT is one of the behavioural intervention techniques developed by Herbert Benson in 1975. BRT is based on the principle of deep breathing and relaxing all the muscles in the body by choosing a word that is meaningful for the individual and focusing on it. This exercise, which has no side effects on patients and can be applied for patients of all age groups, is more widely used because it is a simple and easy-to-learn method compared to other relaxation methods all the muscles in the body by choosing a word that is meaningful for the individual and focusing on it.
  Arms: Intervention

SUMMARY:
The aim of this study is to investigate the effect of Benson Relaxation Exercises on sleep quality in hospitalized patients diagnosed with lung cancer. It is planned to be conducted as a randomized controlled trial.

Hypotheses of the Study H1: The sleep quality of lung cancer patients who undergo Benson relaxation exercises is statistically significantly better than that of patients who do not undergo such exercises.

H2: There is no significant difference in sleep quality between patients who undergo Benson relaxation exercises and those who do not.

DETAILED DESCRIPTION:
This study is planned to be conducted between September 2025 and June 2026 with patients receiving inpatient treatment at the chest ward of a state hospital in Turkey. Patients with lung cancer, pneumonia, type 2 respiratory failure, haemoptysis and tuberculosis receive inpatient treatment at this hospital. A total of 1,787 patients have been treated as inpatients at the hospital in the past year. Patients stay in single rooms. Patients do not engage in any activities other than medical treatment and care.

Participants

The research universe consists of 196 patients diagnosed with lung cancer who are undergoing inpatient treatment at the state hospital's chest clinic. Patients who are unconscious and unable to communicate will be excluded from the research. Randomisation will be applied to the number of patients to be obtained.

In the randomisation phase of the study, Statistical Analysis Software will be used to randomly assign patients. Patients will be randomly assigned to groups using this programme. Patients included in the study will be numbered according to their order of arrival and assigned to the intervention and control groups according to the order in the randomisation list. One of the researchers will be responsible for assigning patients to groups using the Statistical Analysis Software program. This researcher will not participate in the Benson exercises conducted with the patients. Since none of the researchers will know which patients are in the study group, the study will be conducted using a single-blind method. Accordingly, the study is planned to be terminated when a total of 60 patients, including 30 intervention and 30 control groups, are reached.

After reaching the sample size of 60, a power analysis is planned to be performed using the GPower 3.1 programme at a 95% confidence interval.

Sampling Inclusion and Exclusion Criteria:

Inclusion Criteria:

* Be 18 years of age or older,
* Have been diagnosed with lung cancer and be receiving inpatient treatment,
* Be conscious and able to communicate,
* Agree to participate in breathing exercises during the study,
* Score above 5 on the PSQI,
* Have signed the written informed consent form.

Exclusion Criteria:

* Those with additional mental or cognitive disorders,
* Those with physiological barriers to performing breathing exercises,
* Those unable to complete the programme during the study period,
* Those with a PSQI score above 5,
* Those who violate the study protocol,
* Those with an oxygen saturation value below 90,
* Those scoring above 5 on the Visual Pain Scale,
* Those who have previously practised yoga or meditation,
* Patients with haemoptysis
* Patients taking any anxiolytic or hypnotic medication

During the 15 days of Benson relaxation exercise, patients in both the intervention and control groups will not be allowed to perform the exercise if their O2 saturation and pain level changes meet the exclusion criteria.

Measurement

Patient file information , patient identification form , oxygen saturation information , visual analogue scale (VAS) and Pittsburgh Sleep Quality Index (PSQI) will be used to collect data.Patient File Information; this form, developed by researchers, includes questions about the duration of the disease, the stage of the disease, treatment of the disease, the presence of additional mental illness in the patient, whether there are any obstacles to performing breathing exercises, whether the patient has previously practised meditation, the presence of haemoptysis, use of anxiolytic medication, oxygen saturation value, visual pain scale score, and questions regarding the patient's level of consciousness.Patient Identification Form;developed by researchers, this form contains six questions designed to determine sociodemographic characteristics such as age, gender, educational status, employment status, pain, and smoking habits. Oxygen Saturation Information; oxygen saturation refers to the amount of oxygen carried in the blood bound to haemoglobin. In a normal healthy person, PaO2 in the blood is 95 mmHg, and SaO2 is approximately 97%. When arterial oxygen saturation (SaO2) falls below 90%, this is called hypoxemia. SpO₂ 95-100%: Normal, SpO₂ 91-94%: Mild hypoxia, SpO₂ 86-90%: Moderate hypoxia, SpO₂ below 85%: Severe hypoxia .Visual Analogue Scale (VAS); a scale used to determine the intensity and level of pain, consisting of a straight line measuring 10 cm, where '0' indicates no pain and '10' indicates very severe pain. Patients are asked to mark the point on the line that corresponds to the intensity of pain they are feeling. The centimetre equivalent of the marked point is then evaluated as the 'intensity of pain.Pittsburgh Sleep Quality Index - PSQI (The Pittsburgh Sleep Quality Index); the validity and reliability of this scale, developed by Buysse et al. (1989), was established by Ağargün et al. (1996). The PSQI provides a quantitative measurement of sleep quality that helps to define good and poor sleep. The PSQI consists of a total of 24 questions. Nineteen of these questions are self-assessment questions, while five questions are answered by the individual's spouse or a friend. These five questions are used solely for clinical information and are not included in the assessment. Question 19 of the self-assessment questions relates to whether the individual has a roommate or spouse and is not considered in determining the total and component scores of the scale. The self-assessment questions cover various factors related to sleep quality. These include sleep duration, sleep latency (the time it takes to fall asleep), and the frequency and severity of specific sleep-related problems. The 18 scored items are grouped into 7 component scores. Some components consist of a single item, while others are derived from grouping several items. Each item is scored on a scale of 0-3. The sum of the seven component scores yields the total PSQI score. The total score ranges from 0 to 21. A high total scale score indicates poor sleep quality. A total PSQI score of 5 or higher indicates poor sleep quality.

Prosedur

The study plans to use educational booklets containing Benson's application steps to be given to the intervention group. The content of the educational booklets will be created by the researchers. A pilot study is planned with six patients who meet the research criteria and have agreed to participate in the study, in order to assess the clarity of the commands in the data collection forms and the booklet, the adequacy of the time frame, and to obtain patient feedback. Following the pilot study, necessary changes to the data collection forms and educational booklets are planned.Although the length of hospital stay for patients in this study varies depending on their illness and progress in treatment, as a standard practice of the hospital, patients receive treatment in the clinic for an average of three weeks. Therefore, it is planned to apply BRT to the intervention group for two weeks and to conduct a follow-up evaluation in the third week. This exercise, which will be administered once daily to patients in the intervention group during their two-week hospital stay through individual sessions, is planned to be conducted in a quiet room, with each session lasting 20 minutes. The researcher has undergone training in this area and plans to administer the intervention to patients personally.BRT is one of the behavioural intervention techniques developed by Herbert Benson in 1975.BRT is based on the principle of choosing a meaningful word for the individual, focusing on it, taking deep breaths and relaxing all the muscles in the body. This exercise, which has no side effects on patients and can be applied to patients of all age groups, is more widely used than other relaxation methods because it is simple and easy to learn.

The stages of Benson's relaxation exercise are listed below. These stages are given as commands by the practitioner to the person performing the exercise. The exercise lasts an average of 10 to 20 minutes. The commands to be given to the intervention group during the application phase of the study are as follows.

1. Choose a short sentence or word that is meaningful to you and helps you focus your attention. This could be 'health, well-being, abundance' or 'love.'
2. Sit quietly in a comfortable position.
3. Close your eyes.
4. Starting from your feet, slowly move upward toward your muscle groups, relaxing the muscles in your calves, thighs, abdomen, chest, shoulders, neck, and head.
5. Breathe slowly and naturally, and as you exhale, silently repeat your focus word, sound, phrase, or prayer.
6. Adopt a passive attitude. Do not think about whether you are doing it right or wrong. When other thoughts come to mind, tell yourself, 'Everything is fine,' 'I am relaxed, healthy, and energetic,' and calmly focus on your breathing and muscles.
7. Focus on relaxing and letting go until the instructions are finished.
8. Do not get up immediately after the instructions are finished. Continue sitting quietly for one or two minutes to acclimate yourself to your surroundings. Then remove the blindfold from your eyes, slowly open your eyes, and sit for another one or two minutes before getting up. These are the steps involved.

Statistical analysis of the data

The analysis of the data obtained in this study will be performed using the SPSS 26.0 statistical programme. Descriptive data will be presented as mean, frequency, percentage, and standard deviation. Normality tests will be used to evaluate differences in qualitative characteristics between the two groups. Parametric tests will be preferred when the normal distribution assumption is met, and non-parametric tests will be preferred when it is not met. Additionally, independent sample t-tests are planned to be used to examine differences in mean scores between the intervention and control groups (e.g., Pittsburgh Sleep). After the intervention, a covariance analysis (ANCOVA) will be conducted to compare sleep quality scores between the intervention and control groups, and confounding variables (e.g., pre-test scores and group factors) will be controlled for. Additional advanced analyses will be used to eliminate confounding variables. A significance level of p <0.05 will be applied for all statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and over,
* Have been diagnosed with lung cancer and be receiving inpatient treatment,
* Be conscious and able to communicate,
* Agree to participate in breathing exercises during the study,
* Score above 5 on the PSQI,
* Sign a written informed consent form.

Exclusion Criteria:

* Patients under 18 years of age,
* Those with additional mental or cognitive disorders,
* Those with physiological barriers to performing breathing exercises,
* Those unable to complete the programme during the study period,
* Those with a PSQI score above 5,
* Those who violated the study protocol,

  •. Those with an oxygen saturation value below 90,
* Those scoring above 5 on the Visual Pain Scale,
* Those who have previously practised yoga or meditation,
* Patients with haemoptysis,
* Patients taking any anxiolytic or hypnotic medication.

  * During the 15 days of Benson relaxation exercise, patients in both the intervention and control groups will not be allowed to perform the exercise if their O2 saturation and pain level changes meet the exclusion criteria.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Sleep quality-Pittsburg Sleep Quality Index (PSQI) | up to 6 months
  The Pittsburgh Sleep Quality Index (PSQI)

IPD SHARING:
Plan to Share IPD: No